CLINICAL TRIAL: NCT06020547
Title: Cystic Fibrosis in Adults and Frailty
Brief Title: Cystic Fibrosis and Frailtyh What's in Common?
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Graziamaria Corbi, Associate Professor, Federico II University
Other Study IDs: CysFiFRa
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Frailty Syndrome; Cystic Fibrosis
Keywords: functional status; frailty; Cystic Fibrosis; geriatric syndrome
MeSH Terms: conditions — Frailty; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with Cystic Fibrosis: All patients who met the diagnostic criteria for CF, over 18 years old, with pathological sweat chloride levels (chloride >60 mEq/L) and two CFTR mutations were recruited.
  Sweat chloride levels have been tested, and a panel of CFTR mutations screened. The CFTR genotype has been defined through the screening of the most frequent mutations and rearrangements.

SUMMARY:
The goal of this observational study is to assess the main clinical and anamnestic characteristics, and frailty syndrome in an adult Cystic Fibrosis population. The main question it aims to answer is the possible association of the frailty status with the main clinical, therapeutical characteristics, including the genotyping classification of Cystic Fibrosis patients.

DETAILED DESCRIPTION:
Participants will be assessed for the pulmonary status by spirometry (for Forced Expiratory Volume in 1 second [FEV1 - L]; Forced Expiratory Volume in 1 second percent predicted [ppFEV1%]; Forced Vital Capacity [FVC - L]; Forced Vital Capacity percent predicted [FVC %]; Maximal Mid-Expiratory Flow [MMEF]); for the functional status by evaluating the activities of daily living [ADLs], and the instrumental ADLs [IADLs]; and for frailty by the Study of Osteoporotic Fractures [SOF] Index. The height and weight will be also recorded, and Body Mass Index [BMI] calculated as body weight divided by height squared [Kg/m2]. Body weight will be measured in a fasting state in the morning with a mechanical balance.

ELIGIBILITY:
Inclusion Criteria:

* who met the diagnostic criteria for CF,
* over 18 years old,
* pathological sweat chloride levels (chloride >60 mEq/L) and two CFTR mutations

Exclusion Criteria:

* who did not meet the diagnostic criteria for CF
* under 18 years old
* over 18 years old with normal sweat chloride levels (chloride >60 mEq/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population consists of 139 CF patients referred to the Cystic Fibrosis for the Adults Centre of the University Federico II of Naples.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Pre-Frail/Frail Status | through study completion, an average of 1 year
  Frailty has been assessed by the SOF Index

CONTACTS AND LOCATIONS:
Overall Officials: Graziamaria Corbi, MD, PhD, Principal Investigator — Federico II University
Locations (1):
- Cystic Fibrosis for the Adults Centre, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided
the data will be treated as pooled